CLINICAL TRIAL: NCT04042714
Title: An Open-label, Phase II Investigation of TAS-102 in Patients With High Grade, Extrapulmonary Neuroendocrine Carcinoma
Brief Title: TAS-102 in Extrapulmonary Neuroendocrine Carcinoma
Acronym: TAS-102 NEC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted due to low enrollment
Sponsor: Baylor Research Institute (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 019-075; 019-075 (Other: Baylor Scott and White Research Institute)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2020-01

CONDITIONS: High-grade Extra Pulmonary Neuroendocrine Cancer
MeSH Terms: interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: Patients with metastatic high-grade extra pulmonary NEC, who failed front line treatment with a platinum containing regimen, who meets the enrollment criteria will receive TAS-102 as a single agent until either progression or unacceptable toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS-102 (Experimental): Patients will receive TAS-102, Orally, BID for 5 days a week with 2 days rest for 14 days, followed by a 14-day rest treatment cycle. Treatment may continue until disease progresses, intolerable toxicity is developed, or if the patient becomes pregnant or dies.
  Interventions: Drug: All patients- TAS-102

INTERVENTIONS:
Drug: All patients- TAS-102 — Patients will receive TAS-102, Orally, BID for 5 days a week with 2 days rest for 14 days, followed by a 14-day rest treatment cycle. Treatment may continue until disease progresses, intolerable toxicity is developed, or if the patient becomes pregnant or dies.
  Other Names: Trifluridine, Tipiracil

SUMMARY:
The purpose of this study is to test the safety and efficacy of drug, TAS-102 (trifluridine/tipiracil), in patients with extrapulmonary (outside the lung) high-grade neuroendocrine cancer. TAS-102 demonstrated improved survival and tolerability in patients with colorectal cancer and is currently approved by the FDA and marketed under the brand name Lonsurf for the treatment of patients with metastatic colorectal cancer (mCRC). Recently, a study evaluating TAS-102 showed a case of complete remission of high-grade NEC. Given the safety profile of TAS-102 and the remarkable single agent activity in a disease with otherwise dismal outcomes, we hope that TAS-102 may show tolerability and efficacy in neuro-endocrine cancer and propose further exploration in patients with extrapulmonary (outside the lung) high-grade neuroendocrine cancer.

DETAILED DESCRIPTION:
Neuroendocrine tumors are highly prevalent cancer showing heterogeneous array of behaviors. For intermediate/high grade and poorly differentiated neuroendocrine carcinomas (NEC) that occur outside the lung, there is no acceptable standard of care. Most patients are treated with a platinum-based chemotherapy in the front-line setting and evidence for therapies in the second line setting is minimal representing a significant unmet need. However, the response rates have been unsatisfactory with progression-free survival of only 2.3 to 6.2 months, and there is an unmet need for an effective treatment for patients with refractory disease.

TAS-102 is a novel combination medicinal product consisting of a thymidine-based nucleoside analogue (trifluridine; FTD) as the active component and the thymidine phosphorylase inhibitor tipiracil hydrochloride (TPI) that has shown promising activity in phase I trials in patients with solid tumors and phase II in patients with gastric cancer. FTD enters cancer cells, interferes with DNA synthesis, inhibits cell proliferation and inhibit tumor growth. TPI helps FTD sustain its level in cells without degradation by thymidine phosphorylase (Tpase).Thus TAS-102 uses dual approach to inhibit rapid degradation of trifluridine and subsequent tumor growth.

Given the safety profile and efficacy, the study is designed to explore/evaluate efficacy of TAS-102 and identify characteristics of patients who may respond to this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of high grade NEC using WHO criteria as determined by Ki67>20%, poorly differentiated (G3) characteristics, or >20 mitotic figures/10 high-power fields.
* Unknown primary may be included. Suspected extrapulmonary patients with known lung primary will be excluded.
* Prior treatment with a platinum containing regimen
* RECIST 1.1 measurable disease
* Evidence of stage IV, metastatic disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Serum albumin ≥2.5 gm/dL.
* Expected survival ≥3 months.
* Adequate hematologic function as defined by: a) Absolute neutrophil count (ANC) >1500/mm3; b) Platelets ≥75,000/mm3; c) Hemoglobin >8 g/dL (in the absence of red blood transfusion).
* Adequate liver function, as defined by: a) Serum total bilirubin ≤2.5 x ULN mg/dL. b) ALT (SGPT) and AST (SGOT) ≤5 x upper limit of normal (ULN).
* Adequate renal function, as defined by serum creatinine ≤2.0 x ULN, or creatinine clearance ≥30 mL/min
* Females of child bearing potential must agree to use contraception to avoid pregnancy throughout the study.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Evidence of low-grade or well-differentiated features as determined by the investigator.
* Functional neuroendocrine tumors are excluded.
* Known pulmonary primary or small cell lung cancer will be excluded.
* Significant or uncontrolled congestive heart failure (CHF), myocardial infarction or significant ventricular arrhythmias within the last six months.
* Active infection or antibiotics within 48 hours prior to study enrollment, including unexplained fever (temp > 38°C).
* Other severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as: a) Severe impaired lung functions as defined by spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air, b) Uncontrolled diabetes,c) Liver disease such as cirrhosis or severe hepatic impairment, d) Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the integrity of the study.
* Taking other investigational or anti-cancer treatments while participating in this study. Concurrent radiotherapy is allowed provided to non-target lesions. If target lesions have received radiation therapy, progression must have been demonstrated prior to enrollment.
* Prior or concurrent malignancy, except for the following: a) Adequately treated basal cell or squamous cell skin cancer; b) Cervical carcinoma in situ; c) Adequately treated Stage I or II cancer from which the subject is currently in complete remission; d) Or any other cancer from which the subject has been disease-free for 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 24 months
  To assess clinical activity [ORR = Partial response (PR)+Complete response (CR) ] of TAS-102 in patients with metastatic, extra pulmonary high grade NEC

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  To assess OS in patients with metastatic extra pulmonary high grade NEC who received TAS-102 In comparison with historical records.
Progression free survival (PFS) | 24 months
  To assess PFS in patients with metastatic extra pulmonary high grade NEC who received TAS-102 in comparison with historical records

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott and White University Medical Center,, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No